CLINICAL TRIAL: NCT04081727
Title: Zip-Stitch™ for Vaginal Cuff Closure in Laparoscopic Hysterectomy - Safety & Efficacy Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After the second surgery, enrollment was stopped for reasons unrelated to the study design or test article.
Sponsor: ZSX Medical LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QD-PRO-045 Rev002
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Results first posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Laparoscopic Hysterectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Test Article - Zip-stitch Clips (Experimental): Zip-stitch clips for vaginal cuff closure during laparoscopic hysterectomy
  Interventions: Device: Zip-stitch(TM)
- Reference Group - V-Loc Barbed Suture (Other): Will not be comparative against the test article, but will be performed for reference and safety.
  Interventions: Device: Zip-stitch(TM)

INTERVENTIONS:
Device: Zip-stitch(TM) — The assigned intervention is used to close the cuff following colpotomy.

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of the Zip-stitch™ Vaginal Cuff Closure System. This will be primarily done by measuring the frequency of implant passing following system use. Also assessed will be relevant safety and efficacy endpoints as compared to a two-to-one reference group (V-LOC barbed suture).

DETAILED DESCRIPTION:
This is a prospective, blinded, randomized, controlled study to assess the safety and efficacy of the Zip-stitch™ System in maintaining vaginal cuff closure following laparoscopic hysterectomy. Participating subjects will be randomized and evaluated for implant passing, successful cuff closure, healing, adverse events, dyspareunia, and pain. Blinded follow-up will involve in-person visits at one week, six weeks, and six months. There will be an additional unblinded follow-up by telephone at 12 months post operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated Informed Consent Form 2. Stated willingness to comply with all study procedures, including participation in follow-up visits and telephonic follow-up 3. Female 18 years and older 5. Indicated for Laparoscopic Hysterectomy (may include TLH, LAVH, robotic assisted vaginal hysterectomy)

Exclusion Criteria:

1. History of HIV
2. History of Hepatitis C
3. History of diabetes, that in the opinion of the investigator may delay healing
4. Current use of systemic corticosteroids
5. Active infection of genitals, vagina, cervix, uterus or urinary tract
6. Active bacteremia, sepsis or other active systemic infection
7. Presence of Sexually Transmitted Infection (STI)
8. Evidence of pelvic inflammatory disease (PID)
9. Known clotting defects or bleeding disorders
10. Hemoglobin < 8 g/dL
11. Metastatic disease
12. On anticoagulant therapy
13. Participation in another interventional trial
14. Pregnancy
15. Abnormal PAP results that have not been fully evaluated, or in the opinion of the investigator may indicate abnormal vaginal cuff healing
16. Co-morbidities that, in the opinion of the investigator, may indicate risk of abnormal vaginal cuff healing
17. Intra-op: Bowel injury during laparoscopic hysterectomy procedure prior to attempted cuff closure

16. Intra-op: Bladder injury during laparoscopic hysterectomy procedure prior to attempted cuff closure 17. Intra-op: Cases in which surgeon cannot identify adequate tissue along the cuff to apply suture laparoscopically 18. Intra-op: Cases requiring conversion to laparotomy prior to study intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female subjects are eligible to participate in this study as it concerns intervention during laparoscopic hysterectomy.
Enrollment: 2 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O Holtz, M.D., Principal Investigator — Main Line Health
Locations (1):
- Lankenau Medical Center, Wynnewood, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After the second surgery, enrollment was stopped for reasons unrelated to the study design or test article. The study was not resumed, so enrollment was ended with two subjects.
Groups:
- Test Article - Zip-stitch(TM) Clips: Zip-stitch(TM) clips for vaginal cuff closure during laparoscopic hysterectomy
  Zip-stitch(TM): The Zip-stitch™ system is comprised of a handheld applicator and clip loading tool compatible with standard 10mm trocars and laparoscopic surgical equipment as well as a set of bio-absorbable poly p dioxanone (PDO) clips. This system was developed specifically for closure of the vaginal cuff during laparoscopic hysterectomy as a replacement for traditionally cumbersome laparoscopic suture techniques.
- Reference Group - Vicryl Suture: Will not be comparative against the test article, but will be performed for reference and safety.
Period: Overall Study
Arm/Group | Test Article - Zip-stitch(TM) Clips | Reference Group - Vicryl Suture
Started | 2 | 0
As-treated Analysis | 1 | 1
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was stopped after two subjects enrolled
Groups:
- Test Article - Zip-stitch Clips: Zip-stitch clips for vaginal cuff closure during laparoscopic hysterectomy
  The Zip-stitch™ system is comprised of a handheld applicator and clip loading tool compatible with standard 10mm trocars and laparoscopic surgical equipment as well as a set of bio-absorbable poly-p-dioxanone (PDO) clips. This system was developed specifically for closure of the vaginal cuff during laparoscopic hysterectomy as a replacement for traditionally cumbersome laparoscopic suture techniques.
- Reference Group - Vicryl Suture: Will not be compared against the test article, but will be performed for reference and safety.
- Total: Total of all reporting groups
Arm/Group | Test Article - Zip-stitch Clips | Reference Group - Vicryl Suture | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (3) |  | 43 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: inches] | 64.5 (3.5) |  | 64.5 (3.5)
Weight [Mean (Standard Deviation); unit: pounds] | 164.5 (39.5) |  | 164.5 (39.5)

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint - Number of Participants With Implant Passing
Description: Frequency of implant passing following laparoscopic vaginal cuff closure within six weeks
Time Frame: Six-weeks post-operative
Population: Data analyzed "as-treated."
Measure: Count of Participants; unit: Participants
Arm/Group | Test Article - Zip-stitch Clips | Reference Group - VICRYL Suture
Number analyzed (Participants) | 1 | 1
Participants | 0 | 1

2. Primary Outcome: Primary Safety Endpoint - Number of Participants With Vaginal Cuff Dehiscence
Description: Frequency of Vaginal Cuff Dehiscence following laparoscopic vaginal cuff closure.
Time Frame: Six-weeks post-operative
Population: Data analyzed "as treated."
Measure: Count of Participants; unit: Participants
Arm/Group | Test Article - Zip-stitch Clips | Reference Group - Vicryl Suture
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With Successful Vaginal Cuff Closure
Description: Binary, visual surgeon cuff closure evaluation
Time Frame: Performed at one week, six weeks, and six months after surgery; reported here at six weeks
Population: Data analyzed "as treated."
Measure: Count of Participants; unit: Participants
Arm/Group | Test Article - Zip-stitch Clips | Reference Group - Vicryl Suture
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

4. Secondary Outcome: Number of Participants With Vaginal Cuff Healing
Description: Binary, visual surgeon cuff healing evaluation
Time Frame: Performed at one week, six weeks, and six months after surgery; reported here at six weeks
Population: Data analyzed "as treated."
Measure: Count of Participants; unit: Participants
Arm/Group | Test Article - Zip-stitch Clips | Reference Group - Vicryl Suture
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

5. Secondary Outcome: Comparison of Number of Participants With Implant Passing - Test to Reference
Description: Percentage of subjects experiencing implant passing will be compared between test and reference groups
Time Frame: evaluated at six months post-operative
Population: Data analyzed "as treated."
Measure: Count of Participants; unit: Participants
Groups:
- Reference Group - Vicryl Suture: Performed for reference and safety.
Arm/Group | Test Article - Zip-stitch Clips | Reference Group - Vicryl Suture
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

6. Secondary Outcome: Percentage of Participants With Implant Passing Events Determined to Impact Patient Safety
Description: Each reported implant passing event will be evaluated for association with adverse events. Compared as a percentage of patients in the test vs. reference groups.
Time Frame: Evaluated after one week, six week, six month, and twelve month follow-up
Population: Data analyzed "as treated."
Measure: Count of Participants; unit: Participants
Arm/Group | Test Article - Zip-stitch Clips | Reference Group - Vicryl Suture
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

7. Secondary Outcome: Comparison of Incidence of Adverse Events - Test to Reference
Description: Adverse events and serious adverse events will be tabulated for both the test and reference groups.
Time Frame: Evaluated after one week, six week, six month, and twelve month follow-up; reported here for all time
Population: Data analyzed "as treated."
Measure: Count of Participants; unit: Participants
Arm/Group | Test Article - Zip-stitch Clips | Reference Group - Vicryl Suture
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

8. Secondary Outcome: Number of Participants With Non-increase in Dyspareunia at Follow-up
Description: Non-increase in reported individual subject dyspareunia from baseline to follow-up will be compared (test versus reference group) using the relevant sexual discomfort module of the Female Sexual Function Index (FSFI). The FSFI is a validated metric of female sexual function, where lower scores indicate poor sexual function. Non-increase in sexual discomfort will be compared between test and control groups.
Time Frame: Six-months post-operative and again at 12 months post-operative
Population: Data analyzed "as treated."
Measure: Count of Participants; unit: Participants
Arm/Group | Test Article - Zip-stitch Clips | Reference Group - Vicryl Suture
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Non-increase in Pain at Follow-up
Description: Non-increase in reported individual subject pain from baseline to follow-up will be compared (test versus reference group) using an 11-point Numerical Rating Scale, where 0 indicates no pain, and 10 indicates maximum possible pain.
Time Frame: Six-months post-operative and again at 12 months post-operative; count is number of subjects with non-increase
Population: Data analyzed "as treated."
Measure: Count of Participants; unit: Participants
Arm/Group | Test Article - Zip-stitch Clips | Reference Group - Vicryl Suture
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: One year
Description: No differences. As per protocol, adverse events are safety data, and are therefore reported on an "as treated" basis.
Arm/Group | Test Article - Zip-stitch Clips | Reference Group - Vicryl Suture
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Article - Zip-stitch Clips (N=1) | Reference Group - Vicryl Suture (N=1)
Cuff cellulitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) — cellulitis of the vaginal cuff

LIMITATIONS AND CAVEATS:
After the second surgery, enrollment was stopped for reasons unrelated to the study design or test article. The study was not resumed, so enrollment was ended with two subjects. There were not sufficient data to draw meaningful conclusions from the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT04081727/Prot_SAP_000.pdf